CLINICAL TRIAL: NCT02745990
Title: Recombinant Human Erythropoietin Improve Neurodevelopmental Outcomes in Extremely Preterm Infants
Acronym: EPO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Huiqing Sun (Other)
Collaborators: Zhengzhou University (Other); Göteborg University (Other)
Responsible Party: Sponsor-Investigator, Huiqing Sun, Director of preterm infants intensive care unit, Zhengzhou Children's Hospital, China
Organization: Zhengzhou Children's Hospital, China (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CZS-EPO
Record Dates: First submitted 2016-03-16; First posted 2016-04-21 (Estimated); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Developmental Disabilities
Keywords: erythropoietin; preterm; brain injury; cerebral palsy; PVL
MeSH Terms: conditions — Developmental Disabilities; Premature Birth; Brain Injuries; Cerebral Palsy | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EPO group (Experimental): In EPO group, The recombinant human erythropoietin (rhEPO) will be given by 500 U/kg/dose intravenously within 72h after birth, and every other day up to 32 weeks of corrected age.
  Interventions: Drug: Recombinant human erythropoietin
- Normal saline (Placebo Comparator): Normal saline is administered the same volume with EPO, intravenously within 72h after birth, and every other day up to 32 weeks of corrected age.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Recombinant human erythropoietin — rhEPO is administered 500IU/kg, intravenously within 72h after birth, and every other day up to 32 weeks of corrected age.
  Other Names: Epoietin Beta
  Arms: EPO group
Drug: Normal saline — Normal salin is administered the same volume with rhEPO intravenously within 72h after birth, and every other day up to 32 weeks of corrected age..
  Arms: Normal saline

SUMMARY:
In the ELGAN (Extremely Low Gestational Age Newborn) study, abnormal brain structure and function were associated with intermittent or sustained systemic inflammation (ISSI). Since EPO has anti-inflammatory properties in the kidney and in muscle as well as growth/trophic properties. Based on its potential for neuroprotection, the prospective randomized and masked study was designed to determine whether rhEPO （500u/kg) was also effective in improving developmental outcomes for extremely low gestational age newborns.

DETAILED DESCRIPTION:
Exogenous erythropoietin (EPO) is currently used to reduce or prevent the need for red blood cell transfusions in preterm infants. Just two decades ago, erythropoietin (EPO) receptors were first identified in the brain, and astrocytes were found to be capable of synthesizing EPO . Subsequently, it was found that cultured hippocampal and cerebral cortical neurons exposed to EPO were spared some of the glutamate-induced cell death seen in neurons not exposed to EPO. Thus began the concept that EPO protects the brain against adversity. Several follow-up studies of children who had participated in trials of recombinant EPO for the prevention or treatment of anemia, term newborn encephalopathy,or retinopathy of prematurity have also provided evidence of neuroprotective effects.

In the ELGAN (Extremely Low Gestational Age Newborn) study, abnormal brain structure and function were associated with intermittent or sustained systemic inflammation (ISSI) . Since EPO has anti-inflammatory properties in the kidney and in muscle as well as growth/trophic properties, we reasoned that elevated circulating levels might convey information about reduced risk of brain damage in ELGANs.

Although major neurodevelopmental disabilities such as cerebral palsy (CP), mental disabilities, and learning and attention deficits during school age figure prominently in the outcomes of ELBW infants, successful neuroprotective interventions have yet to be developed. Investagators designed a prospective, randomized, masked study to evaluate rhEPO during initial hospitalization and follow up, and hypothesized that rhEPO recipients would receive fewer transfusions during initial hospitalization in extremely preterm infants. Based on its potential for neuroprotection, our study was designed to determine whether rhEPO (500 u/kg) was also effective in improving developmental outcomes for extremely low gestational age newborns.

The neurodevelopmental outcomes of rhEPO in treating extremely preterm infants are not clear. Investigators propose an early-childhood neurodevelopmental follow-up study to compare long-term effects of the rhEPO as measured by, Bayley Scales of Infant Development III. We plan to follow extremely low gestational age children around 24 months' corrected age (CA) who are enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants admitted to NICU wuth gestational age less than 28 weeks
* Age less than 3 days;
* parental informed consent.

Exclusion Criteria:

* Major life-threatening anomalies (brain, cardiac, chromosomal anomalies)
* Hematologic crises such as DIC, or hemolysis due to blood group incompatibilities
* Polycythemia (hematocrit > 65);
* Hypertension
* Seizures
* Congenital infection

Ages: 1 Day to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 440 (Estimated)
Dates: Start 2016-05; Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Mortality | 2 years
  To compare the death rate of EPO and control groups at 2 years old
Incidence of neurological disability | 2 years
  To assess the incidence of neurological disability of EPO and control groups at 2 years old

SECONDARY OUTCOMES:
Incidence of MDI<70 | 2 years
  To compare the incidence of MDI<70 via Bayley Scales of Infant Development between the two groups at 2 years old
Incidence of cerebral palsy | 2 years
  To compare the incidence of cerebral palsy between the two groups at 2 years old
Short-term complicatioins | 3 months
  Retinopathy of prematurity, periventricular leukomalacia,Intraventricular hemorrhage, necrotising enterocolitis and sepsis
Incidence of blindness | 2 years
  To compare the incidence of blindness via visual acuity between the two groups at 2 years old
Incidence of deafness | 2 years
  To compare the incidence of blindness via auditory brainstem response measurements between the two groups at 2 years old
Early blood biomarkers for poor neurological outcomes | 4 weeks
  To investigate early blood biomarkers via multi-omics to predict poor neurological outcomes
Brain imaging biomarkers for poor neurological outcomes | Up to 40 weeks of corrected age
  To investigate Brain imaging biomarkers via MRI to predict poor neurological outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Ligong Hou, BD, Study Director — Zhengzhou Children's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rees S, Harding R, Walker D. The biological basis of injury and neuroprotection in the fetal and neonatal brain. Int J Dev Neurosci. 2011 Oct;29(6):551-63. doi: 10.1016/j.ijdevneu.2011.04.004. Epub 2011 Apr 15. PMID 21527338
- [Result] Korzeniewski SJ, Allred E, Logan JW, Fichorova RN, Engelke S, Kuban KC, O'Shea TM, Paneth N, Holm M, Dammann O, Leviton A; ELGAN study investigators. Elevated endogenous erythropoietin concentrations are associated with increased risk of brain damage in extremely preterm neonates. PLoS One. 2015 Mar 20;10(3):e0115083. doi: 10.1371/journal.pone.0115083. eCollection 2015. PMID 25793991
- [Result] Moore EM, Bellomo R, Nichol AD. Erythropoietin as a novel brain and kidney protective agent. Anaesth Intensive Care. 2011 May;39(3):356-72. doi: 10.1177/0310057X1103900306. PMID 21675055
- [Result] Ohls RK, Kamath-Rayne BD, Christensen RD, Wiedmeier SE, Rosenberg A, Fuller J, Lacy CB, Roohi M, Lambert DK, Burnett JJ, Pruckler B, Peceny H, Cannon DC, Lowe JR. Cognitive outcomes of preterm infants randomized to darbepoetin, erythropoietin, or placebo. Pediatrics. 2014 Jun;133(6):1023-30. doi: 10.1542/peds.2013-4307. Epub 2014 May 12. PMID 24819566
- [Result] Zhu C, Kang W, Xu F, Cheng X, Zhang Z, Jia L, Ji L, Guo X, Xiong H, Simbruner G, Blomgren K, Wang X. Erythropoietin improved neurologic outcomes in newborns with hypoxic-ischemic encephalopathy. Pediatrics. 2009 Aug;124(2):e218-26. doi: 10.1542/peds.2008-3553. Epub 2009 Jul 27. PMID 19651565
- [Result] Brown MS, Eichorst D, Lala-Black B, Gonzalez R. Higher cumulative doses of erythropoietin and developmental outcomes in preterm infants. Pediatrics. 2009 Oct;124(4):e681-7. doi: 10.1542/peds.2008-2701. Epub 2009 Sep 28. PMID 19786428
- [Result] Leviton A, Kuban KC, Allred EN, Fichorova RN, O'Shea TM, Paneth N; ELGAN Study Investigators. Early postnatal blood concentrations of inflammation-related proteins and microcephaly two years later in infants born before the 28th post-menstrual week. Early Hum Dev. 2011 May;87(5):325-30. doi: 10.1016/j.earlhumdev.2011.01.043. Epub 2011 Feb 18. PMID 21334149
- [Result] O'Shea TM, Shah B, Allred EN, Fichorova RN, Kuban KCK, Dammann O, Leviton A; ELGAN Study Investigators. Inflammation-initiating illnesses, inflammation-related proteins, and cognitive impairment in extremely preterm infants. Brain Behav Immun. 2013 Mar;29:104-112. doi: 10.1016/j.bbi.2012.12.012. Epub 2013 Jan 4. PMID 23295265
- [Result] Lee SH, Li C, Lim SW, Ahn KO, Choi BS, Kim YS, Moon IS, Kim J, Bang BK, Yang CW. Attenuation of interstitial inflammation and fibrosis by recombinant human erythropoietin in chronic cyclosporine nephropathy. Am J Nephrol. 2005 Jan-Feb;25(1):64-76. doi: 10.1159/000084275. Epub 2005 Mar 2. PMID 15746540
- [Result] Contaldo C, Lindenblatt N, Elsherbiny A, Hogger DC, Borozadi MK, Vetter ST, Lang KS, Handschin AE, Giovanoli P. Erythropoietin requires endothelial nitric oxide synthase to counteract TNF-[alpha]-induced microcirculatory dysfunction in murine striated muscle. Shock. 2011 Mar;35(3):315-21. doi: 10.1097/SHK.0b013e3181fd0700. PMID 20926979
- [Result] Milne S, McDonald J, Comino EJ. The use of the Bayley Scales of Infant and Toddler Development III with clinical populations: a preliminary exploration. Phys Occup Ther Pediatr. 2012 Feb;32(1):24-33. doi: 10.3109/01942638.2011.592572. Epub 2011 Aug 4. PMID 21812743